CLINICAL TRIAL: NCT07355127
Title: Comparison of the Effects of Open Kinetic Chain and Closed Kinetic Chain Exercises on Balance and Vertical Jump Performance in Sedentary Individuals
Brief Title: Open vs. Closed Kinetic Chain Exercises in Sedentary Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, HAKAN AYDIN, Dr., Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 141/2024
Record Dates: First submitted 2026-01-03; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sedentary Behavior; Exercise Training
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: randomized controlled trial, 3 groups: OKC, CKC, and a control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open Kinetic Chain (OKC) Group (Experimental): Participants were divided into three groups using stratified randomization: OKC Group (n = 22),
  Interventions: Other: Open Kinetic Chain Exercise Program
- Closed Kinetic Chain (CKC) Group (Experimental): Participants were divided into three groups using stratified randomization: CKC Group (n = 22),
  Interventions: Other: Closed Kinetic Chain Exercise Program
- Control Group (No Intervention): Participants were divided into three groups using stratified randomization: Control Group (n = 24),

INTERVENTIONS:
Other: Open Kinetic Chain Exercise Program — Exercise Intervention
  Arms: Open Kinetic Chain (OKC) Group
Other: Closed Kinetic Chain Exercise Program — Exercise Intervention
  Arms: Closed Kinetic Chain (CKC) Group

SUMMARY:
The aim of this study was to compare the effects of Open Kinetic Chain (OKC) and Closed Kinetic Chain (CKC) exercises on dynamic balance, static balance, and vertical jump performance in sedentary individuals.

A total of 68 sedentary individuals voluntarily participated in this randomized controlled trial and were allocated into three groups: OKC, CKC, and a control group. Exercise programs were administered to the OKC and CKC groups for four weeks. Assessments were conducted before and after the exercise intervention. Dynamic balance was evaluated using the Y Balance Test (YBT), static balance using the Flamingo Balance Test (FBT), and vertical jump performance (VJP) using the MyJump2 mobile application.

DETAILED DESCRIPTION:
Purpose: The aim of this study was to compare the effects of Open Kinetic Chain (OKC) and Closed Kinetic Chain (CKC) exercises on dynamic balance, static balance, and vertical jump performance in sedentary individuals.

Methods: A total of 68 sedentary individuals voluntarily participated in this randomized controlled trial and were allocated into three groups: OKC, CKC, and a control group. Exercise programs were administered to the OKC and CKC groups for four weeks. Assessments were conducted before and after the exercise intervention. Dynamic balance was evaluated using the Y Balance Test (YBT), static balance using the Flamingo Balance Test (FBT), and vertical jump performance (VJP) using the MyJump2 mobile application. Data were analyzed using analysis of variance (ANOVA) and the paired-samples t-test.

Keywords: Y Balance Test, Flamingo Balance Test, Vertical Jump Performance, Explosive Power, MyJump2

ELIGIBILITY:
Inclusion Criteria:

* Having a sedentary behavior (Daily average step count less than 5000 in a smartphone application for the last 3 months) [9].
* Being between 18-30 years of age.
* Having no known health problems.

Exclusion Criteria:

* Individuals with chronic diseases.
* Individuals who exercised regularly in the last 6 months.
* Individuals who underwent surgical operations in the last 6 months.

Withdrawal Criteria:

* Individuals who could not comply with the exercise program.
* Individuals who experienced health problems preventing them from exercising.
* Individuals who took a break from the exercise program for more than 5 days.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Dynamic Balance | 4 weeks
  Dynamic balance performance was assessed using the highly reliable Y Balance Test (YBT). This test has no minimum or maximum values. Higher scores indicate better dynamic stability..
Static Balance | 4 weeks
  Static balance performance was assessed using the validated and reliable Flamingo Balance Test (FBT). This test has no minimum or maximum values. Higher scores indicate worse static balance.
Vertical Jump Performance (VJP) | 4 weeks
  VJP assessment was performed using the MyJump2 mobile application, which has a validity rate of 99.3% when compared to force platforms. The minimum score for this test is 0, and there is no maximum score. Higher scores indicate better vertical jump/plyometric performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No